CLINICAL TRIAL: NCT05452460
Title: Effect of Mindfulness Training on Mental Fatigue-Related Impairments of Endurance Performance and Inhibitory Control in Athletes: An Event-Related Potential Study
Brief Title: Mindfulness Training, Mental Fatigue, Endurance Performance and Neurocognitive Functions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan Normal University (Other)
Responsible Party: Principal Investigator, Yu-Kai Chang, Professor, National Taiwan Normal University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PACNL_JT_MF_Intervention
Record Dates: First submitted 2022-07-06; First posted 2022-07-11 (Actual); Results first posted 2025-01-30 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2024-12

CONDITIONS: Mindfulness Training; Neurocognitive Function; Sports Performance; Mental Fatigue
Keywords: Mindfulness Training; Mental Fatigue; Inhibitory Control; Endurance Performance; ERP
MeSH Terms: conditions — Mental Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness training group (Experimental): Participants in the mindfulness training (MT) group will engage in a 60-min session of mindfulness program per week for 8 weeks.
  Interventions: Behavioral: Mindfulness intervention
- Waitlist control group (No Intervention): Participants in the waitlist control group will be required to maintain regular life and routine training. Once the participants in control group finished the whole experiment, they will be invited to participate in the MBPP program for eight weeks.

INTERVENTIONS:
Behavioral: Mindfulness intervention — The mindfulness program called "Mindfulness-based peak performance (MBPP)" will be used in this study. MBPP is a program that consists of eight 60-min training, and a 60-min session weekly for 8-weeks. The MBPP program will include (1) 5 minutes of will start with a brief recap of the preceding session and homework discussion, (2) after which the 5 minutes of a brief story about performance aimed at inducing the learning motivation of the participants; (3) Followed by 20 minutes of a theoretical lecture introducing a new topic and then (4) 25 minutes of mindfulness exercise. (5) Finally, how to apply the mindfulness skills to sports context will be discussed at the end of each session for 5 minutes.
  Arms: Mindfulness training group

SUMMARY:
Mental fatigue has been suggested that would impair neurocognitive functions and sports performance. On the other hand, mindfulness training (MT) seems to as a promising approach to attenuate mental fatigue and counteract its detrimental effect on cognitive functions and sports performance. The purpose of the present study is to examine the effect of MT on behavioral and neuroelectric indices of inhibitory control, and endurance performance in mentally fatigued athletes.

DETAILED DESCRIPTION:
Accumulating research indicates that mental fatigue induced by prolonged cognitive tasks would impair neurocognitive functions and sports performance. Additionally, recent studies demonstrate that inhibitory control and endurance performance are significantly susceptible to detrimental effects of mental fatigue. On the other hand, mindfulness training (MT) has been widely been used to enhance cognitive functions and sports performance in neurocognitive and sports research, which has been considered a promising approach for attenuating mental fatigue and counteracting the detrimental effect of mental fatigue. However, the effect of MT on inhibitory control, endurance performance, and underlying mechanisms in mentally fatigued athletes remain unclear.

Therefore, the purpose of the present study is to examine the effect of MT on behavioral and neuroelectric indices of inhibitory control, and endurance performance in mentally fatigued athletes.

Specifically, the targeted primary outcomes are neurocognitive functions (i.e., reaction time, accuracy and ERPs in Flanker task) and endurance performance (i.e., VO2max & time to exhaustion); The secondary outcomes are changes in dispositional mindfulness, subjective (i.e., scores in visual analog scale)/objective (i.e., reaction time, accuracy in Stroop task) mental fatigue, motivation in tasks, and changes in mood state (i.e., BRUMS-C).

ELIGIBILITY:
Inclusion Criteria:

1. Regular sports training at least 4 hours weekly
2. Normal or corrected-to-normal vision
3. Right-handed

Exclusion Criteria:

1. Physical limitation or injury in lower limbs before and during the study
2. Diagnosed or self-reported neurological disorders (e.g., epilepsy)
3. Diagnosed or self-reported major psychiatric illness (e.g., major depression, schizophrenia)
4. Major previous experience with mindfulness training

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2022-02-17 (Actual); Primary Completion 2023-01-10 (Actual); Study Completion 2023-01-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Kai Chang, PhD, Principal Investigator — National Taiwan Normal University
Locations (1):
- Department of Physical Education and Sport Sciences, National Taiwan Normal University, Taipei, Taiwan

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No participants were excluded from the study before assignment to groups.
Period: Overall Study
Arm/Group | Mindfulness Training Group | Waitlist Control Group
Started | 26 | 27
Completed | 22 | 24
Not Completed | 4 | 3
Not completed — Lost to Follow-up | 3 | 3
Not completed — Did not receive intervention | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mindfulness Training Group | Waitlist Control Group | Total
Number analyzed (Participants) | 26 | 27 | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.08 (1.35) | 20.22 (1.50) | 20.15 (1.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 12
  Male | 19 | 22 | 41
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Sport [Count of Participants; unit: Participants]
  Track & field | 7 | 7 | 14
  Judo | 5 | 7 | 12
  Wrestling | 5 | 6 | 11
  Wushu | 9 | 7 | 16
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 167.5 (6.96) | 168.72 (6.62) | 168.12 (6.75)
Weight [Mean (Standard Deviation); unit: kilograms (kg)] | 71.55 (26.88) | 66.88 (10.01) | 69.17 (20.07)
Education level [Mean (Standard Deviation); unit: years] | 14.35 (1.32) | 14.44 (1.40) | 14.40 (1.35)
Training experience [Mean (Standard Deviation); unit: years] | 8.00 (2.06) | 8.18 (2.65) | 8.10 (2.39)
Working memory [Mean (Standard Deviation); unit: units on a scale] — The Digit-Span Test was used to assess working memory at baseline and to compare cognitive function between groups. The Digit-Span Test included both forward and backward digit spans. The scale for the forward digit span ranges from 0 to 16, while the scale for the backward digit span ranges from 0 to 14. A higher score indicates better verbal working memory.
  units on a scale
    Forward digit span | 14.35 (2.02) | 14.22 (1.55) | 14.28 (1.78)
    Backward digit span | 9.27 (2.75) | 10.22 (2.45) | 9.75 (2.62)

OUTCOME MEASURES:

1. Primary Outcome: Inhibitory Control: Reaction Time
Description: Followed by the manipulation conditions, inhibitory control will be evaluated by a Flanker task (i.e., either mental fatigue condition or control condition). In the Flanker task, participants will be presented with five arrows and will be instructed to respond as quickly and accurately as possible to the direction where the middle arrow is pointing (i.e., left or right). Types of trials are the congruent (i.e., > > > > >) and incongruent (i.e., < < > < <). The reaction time (RT) and accuracy (ACC) of the incongruent trials were calculated as inhibitory control performance, and the difference between conditions was further calculated to represent a mental fatigue-related impairment of inhibitory control in pre-test and post-test.
Time Frame: After 30-minute mental fatigue and control conditions at pre-test and post-test (8 weeks)
Measure: Mean (Standard Deviation); unit: millisecond
Arm/Group | Mindfulness Training Group | Waitlist Control Group
Number analyzed (Participants) | 26 | 27
millisecond
  Condition difference in RT of Flanker task (pre-test) | 10.79 (57.89) | 5.47 (42.72)
  Condition difference in RT of Flanker task (post-test) | 4.11 (19.63) | -0.61 (19.90)
Statistical Analysis 1: Comparison: Mindfulness Training Group vs Waitlist Control Group; Test type: Superiority; p > 0.05, ANCOVA; ANCOVA with post-test condition difference in RT as the outcome, with Group as the factor, and pre-test condition difference in RT as the covariate; Mean Difference (Final Values) = 0.11

2. Primary Outcome: Inhibitory Control: Accuracy
Description: as for outcome 1
Time Frame: After 30-minute mental fatigue and control conditions at pre-test and post-test (8 weeks)
Measure: Mean (Standard Deviation); unit: percentage of correct response
Arm/Group | Mindfulness Training Group | Waitlist Control Group
Number analyzed (Participants) | 26 | 27
percentage of correct response
  Condition difference in ACC of Flanker task (pre-test) | 6.15 (11.79) | 2.32 (11.97)
  Condition difference in ACC of Flanker task (post-test) | 2.60 (6.12) | 2.61 (4.83)
Statistical Analysis 1: Comparison: Mindfulness Training Group vs Waitlist Control Group; Test type: Superiority; p > .05, ANCOVA; ANCOVA with post-test condition difference in ACC the outcome, with Group as the factor, and pre-test condition difference in ACC as the covariate; Mean Difference (Final Values) = 0.18

3. Primary Outcome: ERP: N2
Description: The neuroelectrical activities (i.e., N2, P3) during the Flanker task were recorded and analyzed using the Neuroscan system. The difference in neuroelectrical activities between conditions (i.e., mental fatigue condition & control condition) were calculated as mental fatigue-related impairment in neuroelectrical markers of inhibitory control.
Time Frame: After 30-minute mental fatigue and control conditions at pre-test and post-test (8 weeks)
Measure: Mean (Standard Deviation); unit: μV
Arm/Group | Mindfulness Training Group | Waitlist Control Group
Number analyzed (Participants) | 26 | 27
μV
  Condition difference in N2 amplitude at pre-test (incongruent trial) | -1.27 (3.48) | -1.14 (4.85)
  Condition difference in N2 amplitude at post-test (incongruent trial) | 0.72 (4.07) | 0.18 (2.58)
Statistical Analysis 1: Comparison: Mindfulness Training Group vs Waitlist Control Group; Test type: Superiority; p > 0.05, ANCOVA; ANCOVA with post-test condition difference in N2 the outcome, with Group as the factor, and pre-test condition difference in N2 as the covariate; Mean Difference (Final Values) = 0.32

4. Primary Outcome: ERP: P3
Description: as for outcome 3
Time Frame: After 30-minute mental fatigue and control conditions at pre-test and post-test (8 weeks)
Measure: Mean (Standard Deviation); unit: μV
Arm/Group | Mindfulness Training Group | Waitlist Control Group
Number analyzed (Participants) | 26 | 27
μV
  Condition difference in P3 amplitude at pre-test (incongruent trial) | -0.28 (3.85) | 0.19 (5.23)
  Condition difference in P3 amplitude at post-test (incongruent trial) | 0.78 (6.05) | -0.69 (5.60)
Statistical Analysis 1: Comparison: Mindfulness Training Group vs Waitlist Control Group; Test type: Superiority; p > 0.05, ANCOVA; ANCOVA with post-test condition difference in P3 the outcome, with Group as the factor, and pre-test condition difference in P3 as the covariate; Mean Difference (Final Values) = 0.71

5. Primary Outcome: Endurance Performance: Time to Exhaustion
Description: The graded exercise test (GXT) on treadmill was used to assess participant's endurance performance. Bruce protocol will be adopted in the test. The initial speed and grade of the GXT will be set at 2.74 km/hr with a grade of 10% and increase speed and grade every 3 min until participants are voluntarily exhausted. The time to exhaustion (TTE) was recorded as the endurance performance. The difference in TTE between conditions was further calculated (i.e., control condition minus mental fatigue condition) for both the pre-test and post-test.
Time Frame: After 30-minute mental fatigue and control conditions at pre-test and post-test (8 weeks)
Measure: Mean (Standard Deviation); unit: second
Arm/Group | Mindfulness Training Group | Waitlist Control Group
Number analyzed (Participants) | 26 | 27
second
  Condition difference in TTE at pre-test | 28.50 (32.28) | 23.89 (36.43)
  Condition difference in TTE at post-test | -20.06 (33.54) | 13.15 (34.45)
Statistical Analysis 1: Comparison: Mindfulness Training Group vs Waitlist Control Group; Test type: Superiority; p < 0.01, ANCOVA; ANCOVA with post-test condition difference in TTE the outcome, with Group as the factor, and pre-test condition difference in TTE as the covariate; Mean Difference (Final Values) = 13.35 — [F(1, 52) = 13.35, p = .001, ηp2 = .211]

6. Primary Outcome: Endurance Performance: VO2max
Description: The graded exercise test (GXT) on treadmill was used to assess participant's endurance performance. Bruce protocol will be adopted in the test. The initial speed and grade of the GXT will be set at 2.74 km/hr with a grade of 10% and increase speed and grade every 3 min until participants are voluntarily exhausted. The maximum oxygen consumption (VO2 max) was recorded as the endurance performance. The difference in VO2max between conditions was further calculated (i.e., control condition minus mental fatigue condition) for both the pre-test and post-test.
Time Frame: After 30-minute mental fatigue and control conditions at pre-test and post-test (8 weeks)
Measure: Mean (Standard Deviation); unit: ml/kg/min
Arm/Group | Mindfulness Training Group | Waitlist Control Group
Number analyzed (Participants) | 26 | 27
ml/kg/min
  Condition difference in VO2max at pre-test | 0.86 (4.88) | 0.92 (4.12)
  Condition difference in VO2max at post-test | -0.16 (2.92) | -0.02 (3.62)
Statistical Analysis 1: Comparison: Mindfulness Training Group vs Waitlist Control Group; Test type: Superiority; p > 0.05, ANCOVA; Factor: Group Outcome: Post-test condition difference in VO2max Covariate: Pre-test condition difference in VO2max; Mean Difference (Final Values) = 0.02

7. Secondary Outcome: Subjective Mental Fatigue
Description: Both in the baseline and post-intervention, the visual analog scale for mental fatigue (VAS-MF) was used to assess changes in subjective mental fatigue before and after experimental manipulation. The scale ranges from 0 (not at all mentally fatigued) to 100 (extremely mentally fatigued).
Time Frame: Before, after 30-minute Stroop task and after Flanker task in the mental fatigue and control condition at pre-test and post-test (8 weeks)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness Training Group | Waitlist Control Group
Number analyzed (Participants) | 26 | 27
score on a scale
  VAS score at T1 in pre-test (mental fatigue condition) | 25.19 (11.44) | 24.26 (10.89)
  VAS score at T2 in pre-test (mental fatigue condition) | 47.69 (13.66) | 49.07 (16.06)
  VAS score at T3 in pre-test (mental fatigue condition) | 57.12 (16.01) | 55.56 (22.67)
  VAS score at T1 in pre-test (control condition) | 24.81 (13.38) | 21.30 (11.40)
  VAS score at T2 in pre-test (control condition) | 36.92 (16.00) | 39.26 (11.49)
  VAS score at T3 in pre-test (control condition) | 40.77 (16.89) | 40.19 (13.90)
  VAS score at T1 in post-test (mental fatigue condition) | 22.38 (13.43) | 22.78 (11.06)
  VAS score at T2 in post-test (mental fatigue condition) | 48.50 (13.79) | 50.52 (18.09)
  VAS score at T3 in post-test (mental fatigue condition) | 50.77 (15.56) | 50.78 (18.27)
  VAS score at T1 in post-test (control condition) | 21.08 (12.94) | 24.04 (15.63)
  VAS score at T2 in post-test (control condition) | 36.69 (13.49) | 42.04 (14.27)
  VAS score at T3 in post-test (control condition) | 35.08 (10.62) | 42.07 (12.43)
Statistical Analysis 1: Comparison: Mindfulness Training Group vs Waitlist Control Group; Test type: Superiority; p < 0.01, ANOVA; Four-way mixed-design ANOVA: 2 (GROUP) × 2 (CONDITION) × 3 (ASSESSMENT TIME) × 2 (Experiment Phase); Mean Difference (Final Values) = 38.76

8. Secondary Outcome: Objective Mental Fatigue
Description: Both at baseline and post-intervention, participants completed either a 30-min 100% incongruent version Stroop task (i.e., mental fatigue condition) or a 30-min 100% congruent version Stroop task (i.e., control condition). In the Stroop task, accuracy (ACC) was calculated as an index of objective mental fatigue. It is expressed as a percentage, determined by dividing the number of correct responses by the total number of responses.
Time Frame: Post 30-minute mental fatigue and control condition at pre-test and post-test (8 weeks)
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Mindfulness Training Group | Waitlist Control Group
Number analyzed (Participants) | 26 | 27
percentage
  The ACC of Stroop_Block 1 in pre-test (mental fatigue condition) | 87.09 (9.82) | 88.11 (8.92)
  The ACC of Stroop_Block 2 in pre-test (mental fatigue condition) | 83.77 (1.43) | 85.27 (12.18)
  The ACC of Stroop_Block 3 in pre-test (mental fatigue condition) | 82.54 (13.80) | 86.36 (11.12)
  The ACC of Stroop_Block 4 in pre-test (mental fatigue condition) | 83.72 (13.30) | 85.36 (11.24)
  The ACC of Stroop_Block 5 in pre-test (mental fatigue condition) | 82.94 (16.29) | 82.63 (17.43)
  The ACC of Stroop_Block 1 in pre-test (control condition) | 91.65 (6.10) | 92.63 (5.83)
  The ACC of Stroop_Block 2 in pre-test (control condition) | 89.61 (8.53) | 91.52 (5.47)
  The ACC of Stroop_Block 3 in pre-test (control condition) | 86.92 (12.89) | 90.68 (7.03)
  The ACC of Stroop_Block 4 in pre-test (control condition) | 87.94 (8.77) | 88.96 (9.90)
  The ACC of Stroop_Block 5 in pre-test (control condition) | 86.70 (10.68) | 85.62 (11.96)
  The ACC of Stroop_Block 1 in post-test (mental fatigue condition) | 87.25 (8.13) | 87.77 (10.21)
  The ACC of Stroop_Block 2 in post-test (mental fatigue condition) | 84.69 (9.87) | 85.93 (9.81)
  The ACC of Stroop_Block 3 in post-test (mental fatigue condition) | 83.20 (11.14) | 84.73 (11.75)
  The ACC of Stroop_Block 4 in post-test (mental fatigue condition) | 83.70 (10.92) | 84.41 (10.04)
  The ACC of Stroop_Block 5 in post-test (mental fatigue condition) | 82.06 (13.29) | 84.24 (10.86)
  The ACC of Stroop_Block 1 in post-test (control condition) | 93.21 (5.47) | 94.35 (4.42)
  The ACC of Stroop_Block 2 in post-test (control condition) | 90.84 (7.28) | 91.59 (5.93)
  The ACC of Stroop_Block 3 in post-test (control condition) | 90.85 (6.14) | 91.97 (6.27)
  The ACC of Stroop_Block 4 in post-test (control condition) | 88.81 (7.19) | 90.08 (5.86)
  The ACC of Stroop_Block 5 in post-test (control condition) | 87.41 (8.48) | 88.68 (8.09)
Statistical Analysis 1: Comparison: Mindfulness Training Group vs Waitlist Control Group; Test type: Superiority; p < 0.01, ANOVA — The main effect of the Stroop block on accuracy showed a decrease from the first block to the fifth block; Four-way mixed-design ANOVA: 2 (GROUP) × 2 (CONDITION) × 5 (BLOCK) × 2 (Phase); Mean Difference (Final Values) = 9.21

9. Secondary Outcome: Dispositional Mindfulness
Description: The change in dispositional mindfulness was assessed using the 16-item (5-Likert scale) athlete mindfulness questionnaire (AMQ). The mean score range is between 1-5. Higher mean scores indicate a higher level of dispositional mindfulness.
Time Frame: Baseline (pre-test) and 8 weeks (post-test)
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Mindfulness Training Group: Participants in the mindfulness training (MT) group engaged in a 60-min session of mindfulness program per week for 8 weeks.
  Mindfulness intervention: The mindfulness program called "Mindfulness-based peak performance (MBPP)" was used in this study. MBPP is a program that consists of eight 60-min training, and a 60-min session weekly for 8-weeks. The MBPP program will include (1) 5 minutes of will start with a brief recap of the preceding session and homework discussion, (2) after which the 5 minutes of a brief story about performance aimed at inducing the learning motivation of the participants; (3) Followed by 20 minutes of a theoretical lecture introducing a new topic and then (4) 25 minutes of mindfulness exercise. (5) Finally, how to apply the mindfulness skills to sports context will be discussed at the end of each session for 5 minutes.
- Waitlist Control Group: Participants in the waitlist control group was asked to maintain regular life and routine training. Once the participants in the control group finished the whole experiment, they were invited to participate in the MBPP program for eight weeks.
Arm/Group | Mindfulness Training Group | Waitlist Control Group
Number analyzed (Participants) | 26 | 27
score on a scale
  AMQ score in pre-test | 3.94 (0.59) | 4.04 (0.53)
  AMQ score in post-test | 4.13 (0.55) | 3.87 (0.44)
Statistical Analysis 1: Comparison: Mindfulness Training Group vs Waitlist Control Group; Test type: Superiority; p < 0.05, ANCOVA; Factor: Group Outcome: Post-test mean score Covariate: Pre-test mean score; Mean Difference (Final Values) = 7.07

10. Secondary Outcome: Mood State: Anger
Description: Mood state change was determined by the difference in scores on the Brunel Mood Scale-Chinese (BRUMS-C) between before and after manipulation. The BRUMS-C contains 23 item (5-Likert scale) and is divided into six sub-scales: anger, confusion, depression, fatigue, tension, and vigour. The mean score range is between 0-4. Higher mean scores indicate a higher anger mood.
Time Frame: Before, after 30-minute Stroop task in the mental fatigue and control condition at pre-test and post-test (8 weeks)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness Training Group | Waitlist Control Group
Number analyzed (Participants) | 26 | 27
score on a scale
  Change of anger in pre-mental fatigue condition | 0.13 (0.64) | 0.06 (0.24)
  Change of anger in post-mental fatigue condition | 0.21 (0.52) | 0.05 (0.33)
  Change of anger in pre-control condition | 0.12 (0.38) | 0.37 (0.49)
  Change of anger in post-control condition | -0.04 (0.36) | -0.03 (0.31)
Statistical Analysis 1: Comparison: Mindfulness Training Group vs Waitlist Control Group; Test type: Superiority; p > 0.05, ANCOVA; Factor: Group Outcome: Post-test condition difference in changed anger Covariate: Pre-test condition difference in changed anger; Mean Difference (Final Values) = 1.37

11. Secondary Outcome: Mood State: Confusion
Description: Mood state change was determined by the difference in scores on the Brunel Mood Scale-Chinese (BRUMS-C) between before and after manipulation. The BRUMS-C contains 23 item (5-Likert scale) and is divided into six sub-scales: anger, confusion, depression, fatigue, tension, and vigour. The mean score range is between 0-4. Higher mean scores indicate a higher confusion mood.
Time Frame: Before, after 30-minute Stroop task in the mental fatigue and control condition at pre-test and post-test (8 weeks)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness Training Group | Waitlist Control Group
Number analyzed (Participants) | 26 | 27
score on a scale
  Change of confusion in pre-mental fatigue condition | 0.59 (0.78) | 0.56 (0.75)
  Change of confusion in post-mental fatigue condition | 0.70 (0.63) | 0.50 (0.56)
  Change of confusion in pre-control condition | 0.37 (0.49) | 0.29 (0.54)
  Change of confusion in post-control condition | 0.18 (0.40) | 0.30 (0.56)
Statistical Analysis 1: Comparison: Mindfulness Training Group vs Waitlist Control Group; Test type: Superiority; p > 0.05, ANCOVA; Factor: Group Outcome: Post-test condition difference in changed confusion Covariate: Pre-test condition difference in changed confusion; Mean Difference (Final Values) = 2.73

12. Secondary Outcome: Mood State: Depression
Description: Mood state change was determined by the difference in scores on the Brunel Mood Scale-Chinese (BRUMS-C) between before and after manipulation. The BRUMS-C contains 23 item (5-Likert scale) and is divided into six sub-scales: anger, confusion, depression, fatigue, tension, and vigour. The mean score range is between 0-4. Higher mean scores indicate a higher depression mood.
Time Frame: Before, after 30-minute Stroop task in the mental fatigue and control condition at pre-test and post-test (8 weeks)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness Training Group | Waitlist Control Group
Number analyzed (Participants) | 26 | 27
score on a scale
  Change of depression in pre-mental fatigue condition | 0.07 (0.56) | 0.05 (0.38)
  Change of depression in post-mental fatigue condition | 0.17 (0.50) | 0.14 (0.52)
  Change of depression in pre-control condition | 0.12 (0.38) | -0.01 (0.28)
  Change of depression in post-control condition | -0.01 (0.25) | -0.07 (0.38)
Statistical Analysis 1: Comparison: Mindfulness Training Group vs Waitlist Control Group; Test type: Superiority; p > 0.05, ANCOVA; Factor: Group Outcome: Post-test condition difference in changed depression Covariate: Pre-test condition difference in changed depression; Mean Difference (Final Values) = 0.07

13. Secondary Outcome: Mood State: Fatigue
Description: Mood state change was determined by the difference in scores on the Brunel Mood Scale-Chinese (BRUMS-C) between before and after manipulation. The BRUMS-C contains 23 item (5-Likert scale) and is divided into six sub-scales: anger, confusion, depression, fatigue, tension, and vigour. The mean score range is between 0-4. Higher mean scores indicate a higher fatigue mood.
Time Frame: Before, after 30-minute Stroop task in the mental fatigue and control condition at pre-test and post-test (8 weeks)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness Training Group | Waitlist Control Group
Number analyzed (Participants) | 26 | 27
score on a scale
  Change of fatigue in pre-mental fatigue condition | 1.23 (1.07) | 1.26 (1.00)
  Change of fatigue in post-mental fatigue condition | 1.04 (0.90) | 0.86 (0.85)
  Change of fatigue in pre-control condition | 0.98 (0.93) | 0.78 (0.94)
  Change of fatigue in post-control condition | 0.65 (0.92) | 0.64 (0.81)
Statistical Analysis 1: Comparison: Mindfulness Training Group vs Waitlist Control Group; Test type: Superiority; p > 0.05, ANCOVA; Factor: Group Outcome: Post-test condition difference in changed fatigue Covariate: Pre-test condition difference in changed fatigue; Mean Difference (Final Values) = 0.20

14. Secondary Outcome: Mood State: Tension
Description: Mood state change was determined by the difference in scores on the Brunel Mood Scale-Chinese (BRUMS-C) between before and after manipulation. The BRUMS-C contains 23 item (5-Likert scale) and is divided into six sub-scales: anger, confusion, depression, fatigue, tension, and vigour. The mean score range is between 0-4. Higher mean scores indicate a higher tension mood.
Time Frame: Before, after 30-minute Stroop task in the mental fatigue and control condition at pre-test and post-test (8 weeks)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness Training Group | Waitlist Control Group
Number analyzed (Participants) | 26 | 27
score on a scale
  Change of tension in pre-mental fatigue condition | 0.06 (0.69) | 0.14 (0.43)
  Change of tension in post-mental fatigue condition | 0.20 (0.54) | 0.11 (0.42)
  Change of tension in pre-control condition | 0.07 (0.40) | 0.04 (0.54)
  Change of tension in post-control condition | -0.00 (0.35) | -0.05 (0.41)
Statistical Analysis 1: Comparison: Mindfulness Training Group vs Waitlist Control Group; Test type: Superiority; p > 0.05, ANCOVA; [statistical method as in outcome 11, analysis 1]; Mean Difference (Final Values) = 0.01

15. Secondary Outcome: Mood State: Vigour
Description: Mood state change was determined by the difference in scores on the Brunel Mood Scale-Chinese (BRUMS-C) between before and after manipulation. The BRUMS-C contains 23 item (5-Likert scale) and is divided into six sub-scales: anger, confusion, depression, fatigue, tension, and vigour. The mean score range is between 0-4. Higher mean scores indicate a higher vigor mood.
Time Frame: Before, after 30-minute Stroop task in the mental fatigue and control condition at pre-test and post-test (8 weeks)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness Training Group | Waitlist Control Group
Number analyzed (Participants) | 26 | 27
score on a scale
  Change of vigour in pre-mental fatigue condition | -0.92 (0.78) | -1.05 (0.92)
  Change of vigour in post-mental fatigue condition | -0.74 (0.75) | -0.71 (0.72)
  Change of vigour in pre-control condition | -0.81 (0.78) | -0.85 (0.66)
  Change of vigour in post-control condition | -0.49 (0.71) | -0.68 (0.64)
Statistical Analysis 1: Comparison: Mindfulness Training Group vs Waitlist Control Group; Test type: Superiority; p > 0.05, ANCOVA; [statistical method as in outcome 11, analysis 1]; Mean Difference (Final Values) = 0.66

16. Secondary Outcome: Perception of Effort
Description: During the graded exercise test, the perception of effort will be asked at beginning and every 2.5-min using Borg 6 to 20 scale, until the participant comes to voluntary exhaustion.
Time Frame: every 2.5 minutes during graded exercise test
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Through study completion, up to 1 month post-intervention.
Arm/Group | Mindfulness Training Group | Waitlist Control Group
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/27
Other Adverse Events (participants affected / at risk) | 0/26 | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-12-19): https://cdn.clinicaltrials.gov/large-docs/60/NCT05452460/Prot_SAP_000.pdf